CLINICAL TRIAL: NCT05007340
Title: Interstitial Lung Disease in Systemic Autoimmune Rheumatic Diseases (ILD-SARDs) Registry and Biorepository
Brief Title: ILD-SARDs Registry and Biorepository
Acronym: ILD-SARDs
Status: Recruiting | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: McGill University (Other)
Responsible Party: Principal Investigator, Deborah Assayag, Principal Investigator, MD, MAS, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 2021-7678
Record Dates: First submitted 2021-07-29; First posted 2021-08-16 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Interstitial Lung Disease; Systemic Autoimmune Disease; Rheumatic Diseases; Rheumatic Arthritis; Systemic Sclerosis; Autoimmune Myositis; Systemic Lupus Erythematosus; Usual Interstitial Pneumonia; Nonspecific Interstitial Pneumonia
Keywords: Interstitial Lung Disease; Systemic Autoimmune Disease; Rheumatic Diseases; Rheumatic Arthritis; Systemic Sclerosis; Autoimmune Myositis; Systemic Lupus Erythematosus; Usual Interstitial Pneumonia; Nonspecific Interstitial Pneumonia
MeSH Terms: conditions — Lung Diseases, Interstitial; Rheumatic Diseases; Rheumatic Fever; Scleroderma, Systemic; Lupus Erythematosus, Systemic; Idiopathic Pulmonary Fibrosis | interventions — Blood Specimen Collection; Bronchoalveolar Lavage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — * Blood draws: 40 mL (2-3 tbsp) of blood will be drawn in order to collect DNA, RNA, serum and peripheral blood mononuclear cella (PBMCs).
  * For any other tissues or samples: if the patient's medical care or their participation in a research project involves a biopsy or surgery to remove tissue, the tissue not required for diagnosis (excess tissue) or hospital archives will be included in the biobank. This may include healthy tissue as well as tissue affected by the patient's health condition. The Investigators will not conduct extra procedures in order to obtain samples for the sole purpose of this study and will only operate on what's available. These may include blood samples, skin, lung and muscle biopsies, and bronchoalveolar lavage.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood draws — Blood draws will be performed by personnel that are both qualified and authorized by their employer/institution to perform the procedures. The procedures will be performed with standards expected in the context of clinical care. 40 mL (2-3 tbsp) of blood will be drawn in order to collect DNA, RNA, serum and PBMCs. Blood tubes will be sent to the Bank as per the SOP for patient blood sampling and processing. The blood will be processed, centrifuged and stored by a trained laboratory technician.
Other: Other biological samples to biobank (skin, lung and muscle biopsies; bronchoalveolar lavage (BAL fluid) — If the patient's medical care or their participation in a research project involves a biopsy or surgery to remove tissue, the tissue not required for diagnosis (excess tissue) or hospital archives will be included in the biobank. This may include healthy tissue as well as tissue affected by the patient's health condition. The Investigators will not conduct extra procedures in order to obtain samples for the sole purpose of this study and will only operate on what's available. These may include blood samples, skin, lung and muscle biopsies, and bronchoalveolar lavage, all of which will be obtained from the pathology department.
Other: Clinical data collection — Participant's relevant medical information from medical records, general health questionnaires and clinical assessments. The data includes gender, date of birth, race/ethnicity, habits, height, weight, vital signs, medical history, family history, pregnancy history, imaging data pertinent to ILDs and SARDs, results of routine blood tests, environmental exposures, medication and treatment exposures and adherence, function and quality of life, patient's assessment of their own health, clinical symptoms.
Other: Genetic data/DNA/RNA — Results of the DNA or RNA sequencing, conducted for the Biobank and will be made available to future research; possible single nucleotide polymorphism (SNP) assays (including single SNP, low-plex or microarray-based assays).

SUMMARY:
A complex interaction between demographic, environmental and genetic mechanisms impact the onset, severity and outcome of ILD-SARDs through dysregulation of the immune system and lung pro-biotic pathways. Comorbidity and genetic risk indicate that there are overlapping pathogenic mechanisms among SARDs, some of which underlie ILD in different SARDs.

The purpose of this biobank is to study the clinical, pathological, laboratory, and imaging characteristics of SARDs patients with lung involvement. This will help identify as unique features underlying lung involvement in SARDs. In addition, this may lead to the discovery of novel mechanisms of disease and potentially novel targets of treatment for SARDs patients with lung disease.

DETAILED DESCRIPTION:
1. BACKGROUND AND STUDY RATIONALE: Characterized by immune dysregulation with disrupted self-tolerance, systemic autoimmune rheumatic diseases (SARDs) result in inflammation and auto-antibody formation that cause multi-tissue damage. The prototypic SARDs are rheumatoid arthritis (RA), systemic lupus erythematosus (SLE), systemic sclerosis (SSc) and autoimmune myositis (AIM). The lung is a frequent target of autoimmune-mediated injury in patients with SARDs, and interstitial lung disease (ILD) is a major cause of morbidity and mortality in patients with SARDs. Among patients with SARDs, ILD varies widely in terms of its morphological pattern, time course, severity and the specific immune cells and cytokines that are most responsible for lung damage.

Fundamental clinical questions remain unanswered for understanding diagnosis and management of ILD-SARDs:

1. ILD-SARDs prediction: Which patients with SARDs are likely to develop ILD? In retrospective cohorts of patients with RA, a patient's risk of developing ILD can be predicted by their age, sex and presence of auto-antibodies. How these clinical features interact with possible genetic and environmental risk factors needs to be better established to identify SARDs patients most at risk of developing ILD and to design and test interventions that reduce that risk or delay the onset of clinical manifestations in high-risk patients.
2. ILD-SARDs pathogenesis in humans and preclinical models: Why is there considerable heterogeneity in ILD progression and severity in patients with ILD-SARDs? The fundamental changes that occur in the immune system and lungs of patients with ILD-SARDs are still poorly understood. This is in part due to a lack of appropriate pre-clinical models of ILD-SARDs and lung biopsies from patients with ILD-SARDs. Identifying the biologic processes that promote development of ILD in SARDs patients will let the Investigators use drugs for other ILDs to specific patients with ILD-SARDs and promote the development of new targeted therapies.
3. ILD-SARDs treatment: Which are the best therapies for patients with ILD-SARDs? Few proven treatments for patients with ILD-SARDs exist. Many are proposed based only on case reports in specific SARDs. Positive results from studies of anti-fibrotic agents patients show it is possible to reverse the fibrotic process; yet it is unclear whether some patients with ILD-SARDs could also benefit from this approach as it may interact with the immunosuppressive agents the participants already receive. Addressing this issue is critical to changing the natural course of ILD-SARDs, particularly the symptoms and outcomes most important to patients.

The conduct of many of the related future studies will require access to genetic material, fresh peripheral blood cells, serum and tissue from a phenotypically well characterized group of patients with ILD-SARDs. Access to patients is required for future clinical research projects and participation in potential clinical trials. Furthermore, the ILD-SARDs Registry and Biorepository is similar to registries and biorepositories that have been developed or are being developed in Germany, Australia, the United States and elsewhere in Canada. These similarities will facilitate national and international collaboration and allow establishment of a global collaborative network that is essential for further advancement of ILD-SARDs.

The aforementioned future studies that will benefit from the contributions of this Bank include the identification of cell types, immune modulators and genetic pathways dysregulated in ILD-SARDs patients; pre-clinical in vivo and ex vivo models to assess disease pathobiology and targeted interventions, such as mouse models to assess mechanisms in the initiation and progression of ILD in SARDs, as well as a human ILD-SARDs lung-on-a-chip model to assess and predict treatment effect by evaluation mechanical evolution of the tissue; the ILD-SARDs Patient Preferences study, which consists of the facilitation of focus groups to characterize ILD-SARDs patients' experiences, needs and preferences; and the existing open-label, single arm pilot study of the safety and tolerability of nintedanib in patients with ILD and autoimmune inflammatory myopathy, to assess the effect of nintedanib on the state of activation of AIM patients' blood cells and to define its effect on the immunophenotype of circulating blood cells in patients.

2. OBJECTIVES, HYPOTHESIS AND STUDY QUESTIONS A complex interplay between demographic, environmental and genetic mechanisms impact the onset, severity and outcome of ILD-SARDs through dysregulation of the immune system and lung pro-biotic pathways. Co-morbidity and extensive sharing of genetic risk indicate that there are overlapping pathogenic mechanisms among SARDs, some of which underlie ILD in different SARDs. The multidisciplinary team will examine this hypothesis through the establishment of a prospective registry of patients with ILD-SARDs to be enrolled and followed longitudinally, combined with a biorepository.

3. STUDY METHODS The Investigators will develop a longitudinal clinical registry and biorepository of ILD-SARDs patients. Patient recruitment, informed consent, management, storage of data/samples and all other research activities will be done in accordance with the ILD-SARDs Biobank Management Framework. The ILD-SARDs informed consent forms will be used to obtain participant consent. To estimate recruitment in this cohort, the Investigators reviewed the number of patients seen in the multispecialty ILD-SARDs clinic at the McGill University Health Centre (MUHC) over the last year. The Investigators will recruit an inception cohort for biobanking with annual collection of structured clinical data. Clinical data - including clinical rheumatologic and pulmonary assessment, serology, pulmonary function tests, CT imaging, pathology, current treatments - will be collected at every visit. A biorepository will store biological specimens such as blood cells, serum and DNA/RNA for the cohort members. More specifically, the Investigators will collect whole blood samples at visits as defined above. Those belonging to treatment-naive patients will be sent to Dr. David Langlais' lab at the Inflammation Genomics Lab of the McGill University Genome Centre for single cell RNA sequencing and immunophenotyping. A Standard Operating Process (SOP) for blood sampling, shipping and storage has been developed to detail this process. As for whole blood samples coming from non-treatment-naive-patients, those will be sent to Dr. Gregory Fonseca's lab at the Meakins-Christie Lab at the Royal Victoria Hospital to be processed, and the resulting serum will be biobanked. Moreover, patients with an available bronchoalveolar lavage, lung, skin or muscle biopsy, as well as blood samples will be asked for consent for the study staff to access those samples for the purpose of this research. These samples are essential for the mechanisms established in future studies and will help enable them. The PIs, working under different disciplines, will all equally contribute to the study by identifying eligible participants, having medical oversight and study conduct, having written confirmation of inclusion/exclusion criteria, conducting a physical exam, assessing and signing adverse events (AEs) and serious adverse events (SAEs), providing medical care and follow-up to the participant and reviewing, interpreting and signing lab and other test results. Together, this will allow for a larger number of participants to be identified and followed up in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Must be aged 18 years or older
2. Diagnosis of ILD as confirmed by a chest CT
3. Either a defined SARD, an undifferentiated connective tissue disease or features of autoimmunity without meeting clinical criteria for SARD
4. Patient must be willing to give their informed consent and must be able to understand and follow the required study procedures.

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Incident and prevalent ILD-SARDs cases, treatment-naive or non-treatment-naive, followed at the monthly ILD-SARDs clinic at the MUHC will be offered enrollment into this registry at the time when the participants present for their initial or follow-up clinical visit. According to estimations, the Investigators will recruit 252 patients over the initial 5 years. However, the Investigators plan to recruit as many patients as the Investigators can. ILD-SARDs patients identified in the MUHC Pulmonary Clinic or admitted at the MUHC will also be approached and offered enrollment into the registry. Healthy donors that are sex- and relatively aged-matched are welcome for blood draws.
Sampling Method: Non-Probability Sample
Enrollment: 252 (Estimated)
Dates: Start 2021-08-24 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Rate of death or lung transplant via Connective Tissue Disease (CTD) ILD Physician Baseline Respirology Only Form, and CTD ILD Physician Follow-Up Form | 5 years
  Date and cause of death, date of lung transplantation and type (bilateral, single)
Time to acute exacerbations and hospitalizations via ILD-SARDs Additional AcuteSubacute Respiratory Worsening Form, CTD ILD Physician Baseline Respirology Only Form, and CTD ILD Physician Follow-Up Form | 5 years
  Date of worsening symptoms, admission to hospital required (dates of admission and discharge)
Rate of requirement of interventions during hospital admission via ILD-SARDs Additional AcuteSubacute Respiratory Worsening Form, CTD ILD Physician Baseline Respirology Only Form, and CTD ILD Physician Follow-Up Form | 5 years
  Yes or no questions for required ICU stay, required noninvasive ventilation, required mechanical ventilation, required extracorporeal membrane oxygenation (ECMO), bronchoscopy performed, treatment received
Rate of reasons for worsening symptoms via CTD ILD Physician Baseline Respirology Only Form, and ILD-SARDs Additional AcuteSubacute Respiratory Worsening Form | 5 years
  List of possible reasons for worsening symptoms/exacerbations
Rate of outcome of acute exacerbations and hospitalizations via CTD ILD Physician Baseline Respirology Only Form, and ILD-SARDs Additional AcuteSubacute Respiratory Worsening Form | 5 years
  Evaluation of outcome of acute exacerbations and hospitalizations between resolved, plateau with worse symptoms and death
Patient Global Assessment Questionnaire | 5 years
  To measure quality of life and patient related outcomes, ranging from 0 to 10, and where higher scores mean a worse outcome.
36-Item Short Form Survey (SF-36 v2) | 5 years
  To measure quality of life, ranging from 1 to 3 or 5 depending on the question, and where higher scores can either mean a better or worse outcome, depending on the question.
University of California San Diego Medical Center Pulmonary Rehabilitation Program Shortness-of-Breath Questionnaire (UCSD SOBQ) | 5 years
  To measure patient-related outcomes, specifically with dyspnea, ranging from 0 to 5, where higher scores mean a worse outcome.
Functional Assessment of Chronic Illness Therapy - Dyspnea (FACIT-Dyspnea) Questionnaire | 5 years
  To measure patient-related outcomes, specifically with dyspnea, ranging from "No shortness of breath" to "Severely short of breath", including "I did not do this in the past 7 days" with possibility to indicate reason why.
Patient-Reported Outcomes Measurement Information System 29 (PROMIS-29) Questionnaire | 5 years
  To measure patient-related outcomes, specifically with dyspnea, ranging from 1 to 5, where higher scores can mean a better or worse outcome, depending on the question.
King's Brief Interstitial Lung Disease (KBILD) Questionnaire | 5 years
  To measure patient-related outcomes, specifically with dyspnea, ranging from 1 to 7, where higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Pineau, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Inés Colmegna, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Silvia Vidal, PhD, Principal Investigator — McGill University/Research Institute of the McGill University Health Centre
Locations (1):
- RI-MUHC, Montreal, Quebec, Canada